CLINICAL TRIAL: NCT00817011
Title: Phase 4 Study of Development of Pharmacogenomic Method to Predict Antidepressant Responsiveness
Brief Title: Development of Pharmacogenomic Method to Predict Antidepressant Responsiveness
Acronym: PG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., Ph.D, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-03-012
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Antidepressant Drug Adverse Reaction
Keywords: depression; pharmacogenomics; antidepressant response; biological markers; clinical variables
MeSH Terms: conditions — Depression | interventions — Paroxetine; Nortriptyline; Mirtazapine; Bupropion; Duloxetine Hydrochloride; Trazodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRI treated group (Experimental): SSRI treated group are depressive patients treated with fluoxetine, paroxetine, citalopram or sertraline
  Interventions: Drug: SSRI treated group
- non-SSRI treated group (Active Comparator): non-SSRI treated group are depressive patients treated with venlafaxine, nortriptyline, bupropion, duloxetine, trazodone or mirtazapine
  Interventions: Drug: non-SSRI treated group

INTERVENTIONS:
Drug: SSRI treated group — Antidepressant administration of SSRI class for 6 weeks under therapeutic dose
  Other Names: Other Names:; fluoxetine_Prozac; paroxetine_Paxil, Seroxat; sertraline_Zoloft; citalopram_Celexa
  Arms: SSRI treated group
Drug: non-SSRI treated group — Antidepressant administration of non-SSRI class for 6 weeks under therapeutic dose
  Other Names: venlafaxine_Effexor; nortriptyline_Aventyl, Pamelor, Noritren; mirtazapine_Avanza, Zispin, Remeron; bupropion_amfebutamone, Wellbutrin, Zyban; duloxetine_Cymbalta, Yentreve; trazodone_Desyrel, Beneficat, Deprax
  Arms: non-SSRI treated group

SUMMARY:
The Purpose of this study is to predict antidepressant response in advance using pharmacogenomics and peripheral biological markers in depressed patients.

DETAILED DESCRIPTION:
The difficulties to treat depressed patients are 1)the patients don't respond to antidepressant is about 40% of which, and 2) The time lag is existed until the patients respond to antidepressant and show the treatment effects.

If it is predicted the response of antidepressant in advance, it would be overcome such problems. Drug response generally is known to be related to the individual genetic information and the environmental factors. We are going to investigation about antidepressant response using these approaches.

ELIGIBILITY:
Inclusion Criteria:

1. 25 < age <85
2. major depressed patients satisfied with the diagnosis criteria depression of DSM-IV
3. interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

1. received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
2. potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-04; Primary Completion 2016-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
all pharmacogenetic and biological marker variables cause drug response | 24weeks

SECONDARY OUTCOMES:
all clinical cause drug response | 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea